CLINICAL TRIAL: NCT01515449
Title: Predictors of Poor Outcomes in 1038 Sigma Knees
Status: Completed | Type: Observational
Sponsor: NHS Fife (Other Government)
Collaborators: DePuy International (Industry)
Responsible Party: Principal Investigator, Ivan Brenkel, Consultant Orthopaedic Surgeon, NHS Fife
Other Study IDs: IIS2010002
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the project is to ascertain the pre and intra operative predictors of poor outcomes in total knee replacement.

DETAILED DESCRIPTION:
It is known that surgical outcomes are good in the majority following a Sigma knee at 5 years. 3% have persistent pain. Is it possible to predict these patients? Is it possible to make a determination as to which of the 3 outcome measures ((1) American Knee Society Score; (2) SF12 Oxford 12 and (3) Complications) is most appropriate to use and when is the most appropriate time to use it

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing total knee replacement in Fife

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing total knee replacement in Fife
Sampling Method: Non-Probability Sample
Enrollment: 1038 (Actual)
Dates: Start 1998-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Predictors of poor outcomes using 3 measures | 10 years
  A prospective database was set up in October 1998. Patient details were collected preoperatively, intra operatively and immediately post operatively. Patients are then followed up in a dedicated knee clinic at 6 months, 18 months, 3 years and 5 years. Data such as SF12 and the American Knee Society Score was done at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Fife, Kirkcaldy, Fife, United Kingdom